CLINICAL TRIAL: NCT07377552
Title: Association Analysis of Depression and Asthma: A Retrospective Cross-Sectional and Mendelian Randomization Study
Brief Title: Association Analysis of Depression and Asthma
Status: Not yet recruiting | Type: Observational
Sponsor: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Zhenghua Wu, Principal Investigator, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Other Study IDs: ZWu
Record Dates: First submitted 2025-12-23; First posted 2026-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Depression，Asthma
Keywords: Depression，Asthma，Retrospective Cross-Sectional Study，Mendelian Randomization Study

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Depression Group

SUMMARY:
Main Studies Integrate retrospective studies, observational studies, and Mendelian randomization (MR) study methods to systematically analyze the strength and direction of the association between depression and asthma.

Explore whether a causal relationship exists between depression and asthma, and identify potential confounding factors and effect modifiers.

Secondary Studies Screen for key confounding variables that affect the association between depression and asthma (e.g., age, gender, lifestyle, comorbidities, etc.).

Analyze the correlation between depression and the severity of asthma. Verify the stability of instrumental variables (IVs) and the reliability of causal effects in the MR study.

Key Term Supplementary Explanations Effect modifiers: Factors that alter the strength or direction of the association between an exposure (e.g., depression) and an outcome (e.g., asthma) (e.g., certain genes or medications may modify how depression influences asthma risk).

Instrumental variables (IVs): Genetic variants used in MR studies that are associated with the exposure (e.g., depression-related SNPs) but not directly associated with the outcome (e.g., asthma) except through the exposure, helping to reduce confounding and infer causality.

ELIGIBILITY:
Inclusion Criteria For Retrospective Study

* Age ≥ 18 years old
* Complete medical records, including demographic characteristics (age, gender, ethnicity, etc.), clinical diagnosis information (diagnosis time of depression/asthma, diagnostic basis), treatment plans (medication type, dosage), and follow-up records
* Depression diagnosis conforms to relevant clinical criteria; asthma diagnosis conforms to Guidelines for the Prevention and Treatment of Bronchial Asthma (2020 Edition)

For MR Study (GWAS Data)

* Data have undergone strict quality control
* Study participants are of European ancestry (to reduce population stratification bias)
* Clear division of case group and control group, as well as available sample size information

Exclusion Criteria For Retrospective Study

* Comorbidity with other severe mental illnesses (e.g., schizophrenia, bipolar affective disorder)
* Comorbidity with severe respiratory diseases (e.g., chronic obstructive pulmonary disease [COPD], pulmonary fibrosis, lung cancer)
* Comorbidity with severe organ failure (e.g., heart, liver, or kidney failure)
* Lack of key information in medical records (e.g., diagnosis time, core symptoms, treatment plan)

For MR Study (IVs Screening)

* Single nucleotide polymorphisms (SNPs) with an association significance P-value ≥ 5×10-⁸ with the exposure (depression/asthma)
* SNPs with high linkage disequilibrium (LD, r² ≥ 0.001, distance ≤ 10000 kb)
* SNPs located in coding regions or those that may affect gene expression regulation (at risk of horizontal pleiotropy)
* SNPs with an F-statistic < 10 (at risk of weak instrumental variable bias)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Retrospective Study: Participants aged ≥ 18 years who had complete medical records (including demographic characteristics, clinical diagnosis, treatment plan, and follow-up records) between January 2015 and December 2020. Individuals with comorbid severe mental illnesses, severe respiratory diseases, severe organ failure, or missing key information in medical records were excluded.
  MR Study: Participants of European ancestry, with data sourced from the PGC (Psychiatric Genomics Consortium) major depressive disorder GWAS dataset, and the combined asthma GWAS dataset from UK Biobank and GABRIEL Consortium.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2026-01-31 (Estimated); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Integrate retrospective studies, observational studies, and Mendelian randomization (MR) methods to systematically analyze the strength of the association between depression and asthma. | November 1, 2025 - October 31, 2026
  This study integrates retrospective studies, observational studies and Mendelian randomization (MR) to systematically analyze the association strength between depression and asthma. Retrospective studies provide a basis via Meta-analysis of published data. Prospective observational studies verify conclusions and clarify net association by adjusting confounders. MR infers causal links using GWAS-derived SNPs as instruments, with IVW and tests ensuring reliability. This framework clarifies real association strength and causality, supporting comorbidity research.
Explore whether a causal relationship exists between depression and asthma, and identify potential confounding factors. | November 1, 2025 - October 31, 2026
  This study aims to explore the potential causal relationship between depression and asthma, while identifying key confounding factors. Retrospective and prospective observational studies help screen confounders like smoking, BMI, and comorbidities. Mendelian randomization uses GWAS-derived SNPs as instruments to mitigate confounding and reverse causality, with IVW method and reliability tests. It clarifies causal direction and verifies confounding impacts, laying a foundation for comorbidity intervention.
Screen for key confounding variables that influence the association between depression and asthma. | November 1, 2025 - October 31, 2026
  This study focuses on screening key confounding variables that affect the association between depression and asthma. Based on retrospective and prospective observational data, it identifies factors like smoking, BMI, age, gender, and comorbid chronic diseases. Mental stress, socioeconomic status, and medication use are also evaluated. Mendelian randomization further excludes residual confounding, verifying which variables truly mediate their association, to ensure accurate inference of the intrinsic link between the two conditions.
Analyze the correlation between depression and the severity of asthma. | November 1, 2025 - October 31, 2026
  This study analyzes the correlation between depression and asthma severity. Asthma severity is assessed via clinical indicators like lung function (FEV1), symptom frequency, and acute exacerbation rate. Retrospective and observational data are used to quantify their correlation, adjusting for confounding variables. Mendelian randomization excludes reverse causality and residual confounders, clarifying whether depression correlates with aggravated asthma severity, providing insights for targeted comorbidity management.

SECONDARY OUTCOMES:
Verify the stability of instrumental variables (IVs) in the Mendelian Randomization (MR) study. | November 1, 2025 - October 31, 2026
  This study focuses on verifying the stability of instrumental variables (IVs) in the Mendelian Randomization (MR) analysis. SNPs selected from GWAS as IVs are tested for reliability via multiple approaches: linkage disequilibrium filtering, heterogeneity assessment, and horizontal pleiotropy detection using MR-Egger intercept test. Sensitivity analyses, including leave-one-out and IVW robust models, are conducted to confirm IV stability, ensuring no single SNP biases results and reinforcing the credibility of causal inference.

IPD SHARING:
Plan to Share IPD: No